CLINICAL TRIAL: NCT02258841
Title: Testing an Internet-based Safety Decision Aid for Women Experiencing Intimate Partner Violence
Brief Title: Effectiveness of an Online Safety Tool for Canadian Women Experiencing Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of British Columbia (Other); University of New Brunswick (Other); McMaster University (Other); Johns Hopkins University (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Marilyn Ford-Gilboe, Professor and Women's Health Research Chair in Rural Health, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSREB 105436
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Domestic Violence
Keywords: domestic violence; mental health; safety planning
MeSH Terms: conditions — Psychological Well-Being | interventions — Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized online Safety Decision Aid (Experimental): Setting priorities for safety; Danger Assessment; Personalized Action Plan
  Interventions: Behavioral: Setting Priorities for Safety; Behavioral: Danger Assessment; Behavioral: Personalized Action Plan
- General Online Risk/Safety Information (Active Comparator): General Risk and Safety Information; Basic Emergency Safety Plan
  Interventions: Behavioral: General risk and safety information; Behavioral: Basic Emergency Safety Plan

INTERVENTIONS:
Behavioral: Setting Priorities for Safety — Participants rate the importance of 5 priorities to decision-making about their unsafe relationship by comparing the relative importance of each pair of priorities. Weights for each priority are computed and provided to the woman, along with examples of safety strategies that fit with her top ranked priority.
  Arms: Personalized online Safety Decision Aid
Behavioral: Danger Assessment — Participants complete a calendar to show episodes of physical and/or sexual violence they have experienced in the past 12, along with 20 questions assessing risk of serious or lethal violence. A standardized weighted score is provided, along with a brief explanation about her level of danger and appropriate actions she may take.
  Arms: Personalized online Safety Decision Aid
Behavioral: Personalized Action Plan — Women create a tailored action plan for themselves by selecting strategies from 8 different groups, including those which are recommended to them based on their responses to previous questions.
  Arms: Personalized online Safety Decision Aid
Behavioral: General risk and safety information — Participants receive general information about the importance of priorities in making safety decisions and risk factors for intimate partner violence.
  Arms: General Online Risk/Safety Information
Behavioral: Basic Emergency Safety Plan — Participants are provided with a basic emergency plan including information about local DV resources. The information is not personalized but is consistent with online information which women could find on their own (usual care)
  Arms: General Online Risk/Safety Information

SUMMARY:
The purpose of this study is to assess the effectiveness of an interactive, online safety decision aid among diverse Canadian women who are experiencing intimate partner violence (IPV). The investigators will also explore how the online intervention works, and whether it has different effects for different groups of women.

DETAILED DESCRIPTION:
1 in 3 Canadian women experience IPV in their lifetimes. Over time, chronic stress of living in an abusive relationship has been shown to contribute to depression, anxiety and PTSD. Safety planning to reduce the risk of physical and emotional harm in abusive situations is one of the most widely recommended interventions for women in abusive relationship. However, fewer than 1 in 5 Canadian women access support from violence services to assist them in safety planning. Rural, Aboriginal, racialized, immigrant, sexual minority women and women who prioritize their privacy face particular barriers to accessing information and support for safety planning.

We adapted an interactive, online safety decision aid (SDA) recently developed and tested in the U.S. (Glass and colleagues, 2010) so that it applies to diverse groups of Canadian women, and extends the focus on emotional safety. The tool was revised based on a pilot testing for content and usability with 30 women (15 women who had experienced IPV and 15 service providers/experts). In this study, we test the effectiveness of this new tool, called "I CAN Plan 4 Safety" in a sample of 450 women from 3 provinces (ON, BC, New Brunswick). Women will be randomly assigned to complete either the personalized online safety decision aid (intervention) or an online tool which contains general risk and safety information (usual care control). Both tools are located on a confidential, password protected website. After initial completion of the online tools, they will be asked to login to the websites 3, 6 and 12 months later to complete standard outcome assessments. Women may access the information and resources in the online tools at any time for a 12 month period after they enrol in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 19 years and older,
* English-speaking,
* Living in Ontario, New Brunswick, or British Columbia,
* Reports current physical, sexual or emotional abuse in the context of coercive control from a current or former partner (boyfriend, girlfriend, husband, wife, or intimate/sexual partner)
* Expresses comfort with and access to a safe computer with internet
* Access to safe email and mailing address

Exclusion Criteria:

* Men
* Under 19 years of age
* Cannot read/speak English
* Living outside of the 3 study sites
* Uncomfortable using a computer or internet
* No access to a safe computer with internet
* No access to safe email and mailing address
* Does not report current violence from an intimate partner

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms on the Center for Epidemiologic Studies Depression Scale, Revised | baseline, 12 months
  20 item self-report measure used to measure depressive symptoms in community samples and assess the probability of meeting criteria for major depressive disorder
Changes in PTSD symptomology on the PTSD Checklist (Civilian Version) | baseline, 12 months
  17 item self-report measure of PTSD symptoms designed for use in community samples and to assess probability of meeting DSM-IV diagnostic criterial for PTSD

SECONDARY OUTCOMES:
Changes in Decisional Conflict on the low literacy version of the Decisional Conflict Scale | baseline, immediately post-intervention
  The low literacy version of the Decisional Conflict Scale is an established, self-report measure developed by the Ottawa Patient Decision Aids Research Group.
Changes in use of safety strategies on a Safety Behavior Checklist | baseline, 6 months
  self-report measure of use and helpfulness of strategies to deal with violence, adapted from Goodman et als (2003) Intimate Partner Violence Strategies Index
Changes in use of safety strategies on a Safety Behavior Checklist | baseline, 12 months
  self-report measure of use and helpfulness of strategies to deal with violence, adapted from Goodman et als (2003) Intimate Partner Violence Strategies Index
Change in Mastery on Pearlin's Mastery Scale | baseline, 12 months
changes in self-efficacy for safety planning on investigator developed scales | baseline, 6 months
  2 self-report items which assess self-efficacy in making a safety plan for self and for children on a 100 mm visual analogue scale (range 0-100).
changes in self-efficacy for safety planning on investigator developed scales | baseline, 12 months
  2 self-report items which assess self-efficacy in making a safety plan for self and for children on a 100 mm visual analogue scale (range 0-100).

OTHER OUTCOMES:
Severity of violence on the Composite Abuse Scale | baseline, 6, 12 months
  30 item validated measure of severity of intimate partner violence
Social support on the Medical Outcomes Study Social Support Survey | baseline, 3, 6, 12 months
  5 item self-report measure of perceived social support, adapted by McCarrier et al (2011) from the MOS-SS scale
Helpfulness of the online tool to decision making on the Preparation for Decision making scale | immediately post-intervention, 6, 12 months
  10 item self-report measure of helpfulness of the online tool, adapted to IPV context by Glass et al (2010) from the standardized measure developed by the Ottawa Patient Decision Aids Research Group.
Coercive control on the Women's Experiences of Battering Scale (WEB) | baseline, 3, 6, 12 months
  10 item self-report measure of women's responses to partner violence which is a proxy for current level of coercive control

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Ford-Gilboe, PhD, Principal Investigator — Western University
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of New Brunswick, Fredericton, New Brunswick
  - Western University, London, Ontario

REFERENCES:
- [Derived] Ford-Gilboe M, Varcoe C, Scott-Storey K, Perrin N, Wuest J, Wathen CN, Case J, Glass N. Longitudinal impacts of an online safety and health intervention for women experiencing intimate partner violence: randomized controlled trial. BMC Public Health. 2020 Feb 26;20(1):260. doi: 10.1186/s12889-020-8152-8. PMID 32098633
- [Derived] Ford-Gilboe M, Varcoe C, Scott-Storey K, Wuest J, Case J, Currie LM, Glass N, Hodgins M, MacMillan H, Perrin N, Wathen CN. A tailored online safety and health intervention for women experiencing intimate partner violence: the iCAN Plan 4 Safety randomized controlled trial protocol. BMC Public Health. 2017 Mar 21;17(1):273. doi: 10.1186/s12889-017-4143-9. PMID 28327116
- See also: Study Home page. Click here for more information about the iCAN Plan 4 Safety. — http://www.icanplan4safety.ca/index.html